CLINICAL TRIAL: NCT04290728
Title: Effect of High-flow Nasal Oxygenation on Safe Apnea Time in Children With Open Mouth
Brief Title: High-flow Nasal Oxygenation for Open Mouth
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in the study plan
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1910-091-1071
Record Dates: First submitted 2020-02-24; First posted 2020-03-02 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Anesthesia, General; Apnea
Keywords: High-flow nasal cannula; Preoxygenation; Apnea time; General anesthesia
MeSH Terms: conditions — Apnea | interventions — N(6)-2-(4-aminophenyl)ethyladenosine

STUDY DESIGN:
Intervention Model Description: Randomized, controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- High flow (Experimental): Apply high-flow nasal oxygenation during apnea with open mouth after adequate preoxygenation. Resume bag-mask ventilation when pulse oximetry drops to 92% or pre-set apnea time has expired.
  Interventions: Device: Apnea with high-flow nasal cannula
- Control (Active Comparator): Apply nothing during apnea with open mouth after adequate preoxygenation. Resume bag-mask ventilation when pulse oximetry drops to 92% or pre-set apnea time has expired.
  Interventions: Other: Apnea

INTERVENTIONS:
Device: Apnea with high-flow nasal cannula — Application of oxygenation with high-flow nasal cannula with a rate of 2L/kg/min
  Other Names: Airvo 2
  Arms: High flow
Other: Apnea — Apnea without any application of oxygenation
  Arms: Control

SUMMARY:
This study aims to evaluate the effect of high-flow nasal oxygenation on safe apnea time for children undergoing general anesthesia, with their mouth open.

DETAILED DESCRIPTION:
Oxygenation via high-flow nasal cannula is gaining popularity in various clinical settings. It is known to increase apnea time for apneic patients including children. However, high-flow nasal cannula is known to be ineffective when the patient's mouth is kept open.

When trying to intubate the patient during induction of anesthesia, the patient should be apneic with administration of neuromuscular blocking agent, and the mouth should be open for introduction of laryngoscope.

We designed a prospective randomized controlled study to evaluate the effect of high-flow nasal oxygenation in the aforementioned setting for trying to intubate the patient.

ELIGIBILITY:
Inclusion Criteria:

* Children younger than 11 years old scheduled to undergo surgery under general anesthesia, with American Society of Anesthesiologists Physical Status 1 or 2.

Exclusion Criteria:

* Refusal to enrollment from one or more of legal guardians of the patient
* Children who are planned to use supraglottic airway device
* Children with upper respiratory tract infection or pulmonary interstitial disease
* Preterm babies under 40 weeks of postconceptual age
* Children who are expected to have difficult airway for bag-mask ventilation

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Apnea time | Elapsed time starting from discontinuation of oxygen to the time point that pulse oximetry first reaches 92% (not to exceed 520 seconds)
  Time required for pulse oximetry to drop to 92% after start of apnea

SECONDARY OUTCOMES:
End-tidal carbon dioxide | Procedure (From induction of anesthesia to end of anesthesia)
  End-tidal carbon dioxide partial pressure during anesthesia
Pulse oximetry | Procedure (From induction of anesthesia to end of anesthesia)
  Pulse oximetry during anesthesia
Non-invasive blood pressure | Procedure (From induction of anesthesia to end of anesthesia)
  Non-invasive blood pressure measured from forearm or leg
Oxygen reserve index | Procedure (From induction of anesthesia to end of anesthesia)
  Oxygen reserve index measured from finger or toe
Time to 100% | Elapsed time starting from re-start of bag-mask ventilation at the end of apnea period to the time point that pulse oximetry first reaches 100% (estimated less than 2 minutes)
  Elapsed time from re-start of bag-mask ventilation to recovery of pulse oximetry of 100% after apnea
Minimum value of pulse oximetry | Procedure (From induction of anesthesia to end of anesthesia)
  Minimum value of pulse oximetry after re-start of bag-mask ventilation after apnea
1st value of end-tidal carbon dioxide | At expiration of the first manual ventilation after the end of the apnea period (less than 520 seconds after start of apnea period)
  First measured value of end-tidal carbon dioxide partial pressure after re-start of bag-mask ventilation after apnea

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fiadjoe JE, Nishisaki A, Jagannathan N, Hunyady AI, Greenberg RS, Reynolds PI, Matuszczak ME, Rehman MA, Polaner DM, Szmuk P, Nadkarni VM, McGowan FX Jr, Litman RS, Kovatsis PG. Airway management complications in children with difficult tracheal intubation from the Pediatric Difficult Intubation (PeDI) registry: a prospective cohort analysis. Lancet Respir Med. 2016 Jan;4(1):37-48. doi: 10.1016/S2213-2600(15)00508-1. Epub 2015 Dec 17. PMID 26705976
- [Background] Frei FJ, Ummenhofer W. Difficult intubation in paediatrics. Paediatr Anaesth. 1996;6(4):251-63. doi: 10.1111/j.1460-9592.1996.tb00447.x. No abstract available. PMID 8827740
- [Background] Schibler A, Hall GL, Businger F, Reinmann B, Wildhaber JH, Cernelc M, Frey U. Measurement of lung volume and ventilation distribution with an ultrasonic flow meter in healthy infants. Eur Respir J. 2002 Oct;20(4):912-8. doi: 10.1183/09031936.02.00226002. PMID 12412683
- [Background] King W, Petrillo T, Pettignano R. Enteral nutrition and cardiovascular medications in the pediatric intensive care unit. JPEN J Parenter Enteral Nutr. 2004 Sep-Oct;28(5):334-8. doi: 10.1177/0148607104028005334. PMID 15449573
- [Background] Schibler A, Yuill M, Parsley C, Pham T, Gilshenan K, Dakin C. Regional ventilation distribution in non-sedated spontaneously breathing newborns and adults is not different. Pediatr Pulmonol. 2009 Sep;44(9):851-8. doi: 10.1002/ppul.21000. PMID 19672959
- [Background] Schibler A, Henning R. Positive end-expiratory pressure and ventilation inhomogeneity in mechanically ventilated children. Pediatr Crit Care Med. 2002 Apr;3(2):124-128. doi: 10.1097/00130478-200204000-00006. PMID 12780980
- [Background] Erb T, Marsch SC, Hampl KF, Frei FJ. Teaching the use of fiberoptic intubation for children older than two years of age. Anesth Analg. 1997 Nov;85(5):1037-41. doi: 10.1097/00000539-199711000-00013. PMID 9356095
- [Background] Mir F, Patel A, Iqbal R, Cecconi M, Nouraei SA. A randomised controlled trial comparing transnasal humidified rapid insufflation ventilatory exchange (THRIVE) pre-oxygenation with facemask pre-oxygenation in patients undergoing rapid sequence induction of anaesthesia. Anaesthesia. 2017 Apr;72(4):439-443. doi: 10.1111/anae.13799. Epub 2016 Dec 30. PMID 28035669
- [Background] Lodenius A, Piehl J, Ostlund A, Ullman J, Jonsson Fagerlund M. Transnasal humidified rapid-insufflation ventilatory exchange (THRIVE) vs. facemask breathing pre-oxygenation for rapid sequence induction in adults: a prospective randomised non-blinded clinical trial. Anaesthesia. 2018 May;73(5):564-571. doi: 10.1111/anae.14215. Epub 2018 Jan 13. PMID 29330853
- [Background] Humphreys S, Lee-Archer P, Reyne G, Long D, Williams T, Schibler A. Transnasal humidified rapid-insufflation ventilatory exchange (THRIVE) in children: a randomized controlled trial. Br J Anaesth. 2017 Feb;118(2):232-238. doi: 10.1093/bja/aew401. PMID 28100527
- [Background] Lyons C, Callaghan M. Uses and mechanisms of apnoeic oxygenation: a narrative review. Anaesthesia. 2019 Apr;74(4):497-507. doi: 10.1111/anae.14565. Epub 2019 Feb 19. PMID 30784037
- [Background] Wettstein RB, Shelledy DC, Peters JI. Delivered oxygen concentrations using low-flow and high-flow nasal cannulas. Respir Care. 2005 May;50(5):604-9. PMID 15871753
- [Background] Parke R, McGuinness S, Eccleston M. Nasal high-flow therapy delivers low level positive airway pressure. Br J Anaesth. 2009 Dec;103(6):886-90. doi: 10.1093/bja/aep280. Epub 2009 Oct 20. PMID 19846404